CLINICAL TRIAL: NCT01725022
Title: A Controlled Study of Stem Cell Transplantation Medical Home Care Compared to Standard Hospital Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00032263
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Hematologic Malignancies
Keywords: stem cell transplant; bowel microbiota; home care
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Home Care (Experimental): This is the arm for patients who receive their transplant care in their homes.
  Interventions: Other: Home Care
- Hospital Care (No Intervention): Standard of care for stem cell transplant recipients where the aftercare is done in hospital.
- Clinic Care (No Intervention): Standard of care for stem cell transplant recipients who live at home but receive aftercare in the daily outpatient clinic.

INTERVENTIONS:
Other: Home Care — This is the interventional arm where patients receive the transplant care in their homes.
  Arms: Home Care

SUMMARY:
The primary goal with this study is to document whether patients can maintain their normal bowel microbiota by staying at home compared to those who live at home but are treated in clinic, and those who are treated in the hospital. In addition, the investigators would predict that the quality of life will be higher for those patients treated at the medical home compared to those that stay at the hospital. The investigators also predict that the costs associated with this approach will be significantly lower compared to hospitalized patients. Finally, the investigators propose that the treatment related morbidities and mortality will not be different between the two groups.

DETAILED DESCRIPTION:
Subjects enrolled in the medical home arm and those serving as concurrent controls will have the following studies:

1. Stool collection for analysis at time 0 (prior to preparatory regimen) and then weekly for the first four weeks, at day 60 and 100.
2. The PG-SGA, FACT-BMT and other patient-reported symptom instruments will be collected weekly for the first 4 weeks, at day 60, 100 and patients will be required to complete a daily food diary.
3. Other assessments for toxicities or GVHD will proceed as per current standard of care, for a total blood draw amount of 100 mls from home care subjects and concurrent controls.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a hematopoietic stem cell transplant for any cancer or non-cancer illness from any autologous, related or unrelated donor source including bone marrow, peripheral blood progenitor cell, or umbilical cord blood
2. Age 18-80 years of age
3. Karnofsky Performance Scale (KPS) > 80
4. A home that is deemed, upon inspection, in suitable condition to serve as a medical home, within a 90-minute driving distance of Duke (home care group only)

Exclusion Criteria:

1. Lack of a caregiver
2. Pregnant women (It is standard of care to assess for pregnancy for all females of child-bearing potential with a serum beta human chorionic gonadotropin (HCG) test within 7 days of starting the preparative regimen prior to transplant. No additional research pregnancy testing will occur.)
3. Patients with a documented active infection prior to starting their preparative regimen. This includes grade 3 or higher viral, bacterial, or fungal infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-02; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Bowel Microbiota | 100 days
  The bowel microbiota before and during the first 100 days.

SECONDARY OUTCOMES:
Nutritional status using the PG-SGA assessment tool | 100 days
  The assessment tool to capture overall nutritional status will be the Patient Generated Subjective Global Assessment (PG-SGA) which has been validated in other cancer patients.
Incidence of acute Graft Versus Host Disease (GVHD) | 100 days
  All incidences of Grade II-IV GVHD will be quantified.
Treatment related morbidities and mortalities | 100 Days
  Both treatment related morbidities and mortalities will be quantified.
Quality Of Life Assessment (QOL) | 100 Days
  The QOL assessment will utilize the FACT-BMT (Functional Assessment of Cancer Therapy Bone Marrow Transplant) assessment tool as well as other patient-reported symptom instruments to capture the patient reported experience.
Costs of care | 100 Days
  The mean, median and range of costs will be compared in the three arms.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Chao, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States